CLINICAL TRIAL: NCT06199713
Title: Correlation Between Early Interval 18F-Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography (PET/CT) and Circulating Tumor DNA (ctDNA) in Advanced Melanoma Patients Treated With Immune Checkpoint Inhibitors
Brief Title: Correlating Early FDG PET/CT and ctDNA in Immune Checkpoint Inhibitor (ICI)-Treated Melanoma Patients
Status: Recruiting | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-1089; UW23077 (Other: UWCCC); A534260 (Other: UW Madison); Protocol Version 2/12/2024 (Other: UW Madison); NCI-2023-11059 (Registry Identifier: NCI Trial ID)
Record Dates: First submitted 2023-12-27; First posted 2024-01-10 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Melanoma; Melanoma Stage III; Melanoma Stage IV; Unresectable Melanoma
Keywords: circulating tumor DNA; FDG; ICI
MeSH Terms: conditions — Melanoma | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Advanced Melanoma Patients with Immune Checkpoint Inhibitors
  Interventions: Diagnostic Test: 18F-Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography

INTERVENTIONS:
Diagnostic Test: 18F-Fluorodeoxyglucose Positron Emission Tomography/Computed Tomography — research scan 3-4 weeks after start of immunotherapy
  Other Names: 18F-FDG PET/CT

SUMMARY:
The purpose of this research study is to determine if analysis of PET/CT scans and testing of blood samples in people with melanoma that has spread in their body can help researchers determine which patients are more or less likely to respond to immunotherapy and are more or less likely to have side effects. 24 participants will be enrolled and be on study until approximately 4 weeks after their first dose of Immune Checkpoint Inhibitor therapy.

DETAILED DESCRIPTION:
This is a pilot, prospective, observational study to estimate the degree to which baseline and early interval 18F-FDG PET/CT imaging within 3-4 weeks of ICI therapy initiation can accurately correlate with ctDNA level trends, predict clinical response, onset of immune-related adverse events, and survival outcomes in advanced stage melanoma patients.

Primary Objective

• To determine if early interval response assessment with 18F-FDG PET/CT during initial treatment with ICI therapy at 3-4 weeks correlates with ctDNA level changes in advanced melanoma patients.

Secondary Objectives

* To determine if early interval response assessment with 18F-FDG PET/CT during initial treatment with ICI therapy at 3-4 weeks predicts clinical efficacy at standard disease assessment time points in advanced melanoma patients.
* To assess if early interval response assessment with 18F-FDG PET/CT predicts development of clinical irAEs in advanced melanoma patients.
* To assess if early interval response assessment with 18F-FDG PET/CT and ctDNA level predicts progression-free survival (PFS) in advanced melanoma patients.
* To assess if early interval response assessment with 18F-FDG PET/CT and ctDNA level predicts overall survival (OS) in advanced melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Willing to provide informed consent.
* Must have an advanced stage III or stage IV melanoma diagnosis for which treatment with ipilimumab, nivolumab, and/or pembrolizumab, either alone or in combination with other ICI therapy, is planned.
* Must be planning to participate in Signatera™ (ctDNA level) monitoring with standard of care laboratory testing routinely obtained for treatment with ICI therapy.
* Individuals at least 18 years of age.
* Women of childbearing potential must be willing to use effective contraception as discussed with their oncologist while participating in this study.
* Willing to comply with all study procedures and be available for the duration of the study.

Exclusion Criteria:

* Not able to receive treatment with ICI therapy
* Use of investigational drugs, biologics, or devices within 30 days prior to enrollment.
* Women who are pregnant, lactating, or planning on becoming pregnant during the study.
* Not suitable for study participation due to other reasons at the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 24 participants with advanced stage III or stage IV melanoma with measurable disease who are deemed appropriate for treatment with ICI therapy.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Change in ctDNA level from baseline to 3-4 week after the start of therapy | baseline to 3-4 weeks after start of therapy (up to 5 weeks on study)
  ctDNA level is monitored per standard of care in this population, data from chart review.
Change in 18F-FDG PET/CT response from baseline to 3-4 week after the start of therapy | baseline to 3-4 weeks after start of therapy (up to 5 weeks on study)
  Lesion-level and patient-level 18F-FDG PET/CT response assessment at baseline and at 3-4 weeks after starting ICI therapy reported as SUV max.
Correlation between ctDNA level change and 18F-FDG PET/CT response from baseline to 3-4 week after the start of therapy | baseline to 3-4 weeks after start of therapy (up to 5 weeks on study)
  Correlate lesion-level and patient-level 18F-FDG PET/CT response assessment at baseline and at 3-4 weeks after starting ICI therapy with quantitative changes in ctDNA levels at baseline and at 3-4 weeks after starting ICI therapy. Pearson's or Rank's correlation coefficient will be used to measure the baseline measures for ctDNA level trends and PET/CT responses and for those measurements at 3-4 weeks.
Diagnostic Accuracy of ctDNA level trend and PET/CT imaging for predicting growth inhibition as measured by Area under the Curve | baseline to 3-4 weeks after start of therapy (up to 5 weeks on study)
  Receiver-operator curve analysis will be performed to determine the diagnostic accuracy of ctDNA level trend and PET/CT imaging for predicting growth inhibition (area under the curve).

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 12 months after the first ICI dose (approximately 1 year on study)
  Correlate lesion-level and patient-level 18F-FDG PET/CT treatment response assessment at baseline and at 3-4 weeks after starting ICI therapy with clinical response evaluations (RECIST, PERCIST, PECRIT, iRECIST, irRECIST) at 3, 6, 9, and 12 months after the first ICI dose. ORR is Partial Response (PR) plus Complete Response (CR).
Disease Control Rate (DCR) | up to 12 months after the first ICI dose (approximately 1 year on study)
  Correlate lesion-level and patient-level 18F-FDG PET/CT treatment response assessment at baseline and at 3-4 weeks after starting ICI therapy with clinical response evaluations (RECIST, PERCIST, PECRIT, iRECIST, irRECIST) at 3, 6, 9, and 12 months after the first ICI dose. DCR is Stable Disease (SD) plus PR plus CR.
Change in Standard Uptake Value (SUV) metrics with onset of Immune Related Adverse Events (irAE) | up to 12 months after the first ICI dose (approximately 1 year on study)
  Correlate organ-level FDG uptake and changes from the baseline and early 18F-FDG PET/CT assessment with onset of first, second, and third symptomatic irAE per CTCAE v5.0
Progression Free Survival (PFS) | up to 3 years after the first ICI dose (approximately 3 years on study)
  PFS will be summarized using Kaplan-Meier estimates of the median survival times. Point estimates as well as 95% confidence intervals will be provided
Correlation Coefficient for 18F-FDG PET/CT response at 3-4 weeks after the start of therapy and PFS | up to 3 years after the first ICI dose (approximately 3 years on study)
  Correlate early 18F-FDG PET/CT treatment response with Progression Free Survival (PFS) as measured from the date of initiation of ICI treatment until the criteria for disease progression is met as defined by RECIST, PECRIT, or death occurs.
Correlation Coefficient for ctDNA level at 3-4 weeks after the start of therapy and PFS | up to 3 years after the first ICI dose (approximately 3 years on study)
  Correlate early ctDNA level trends with Progression Free Survival (PFS) as measured from the date of initiation of ICI treatment until the criteria for disease progression is met as defined by RECIST, PECRIT, or death occurs.
Overall Survival (OS) | up to 3 years after the first ICI dose (approximately 3 years on study)
  OS will be summarized using Kaplan-Meier estimates of the median survival times. Point estimates as well as 95% confidence intervals will be provided
Correlation Coefficient for 18F-FDG PET/CT response at 3-4 weeks after the start of therapy and OS | up to 3 years after the first ICI dose (approximately 3 years on study)
  Correlate early 18F-FDG PET/CT response assessment with Overall Survival (OS) as measured from the date of initiation of ICI treatment until date of death from any cause.
Correlation Coefficient for ctDNA level at 3-4 weeks after the start of therapy and OS | up to 3 years after the first ICI dose (approximately 3 years on study)
  Correlate early ctDNA level trends with Overall Survival (OS) as measured from the date of initiation of ICI treatment until date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ma, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospitals and Clinics (UWHC), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No